CLINICAL TRIAL: NCT04306640
Title: Demonstration of Autonomic Nervous Function and Cervical Sensorimotor Control After Cervical Lordosis Rehabilitation: A Randomized-controlled Trial
Brief Title: Impact of Cervical Lordosis Rehabilitation on Autonomic Nervous Function and Cervical Sensorimotor Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Associate professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Sharjah
Record Dates: First submitted 2020-03-08; First posted 2020-03-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Chronic Nonspecific Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): the intervention group will receive the denneroll cervical traction orthotic in an attempt to improve the altered sagittal cervical spine alignment (AHT and ARA C2-C7).
  Interventions: Other: Sagittal Cervical Posture Corrective Orthotic Device
- Control group (Active Comparator): Both the intervention group and the control group will complete a multimodal program of 10 weeks consisting of myofascial release, thoracic spine mobilization and manipulations, and physical pain relief methods.
  Interventions: Other: Sagittal Cervical Posture Corrective Orthotic Device

INTERVENTIONS:
Other: Sagittal Cervical Posture Corrective Orthotic Device — The subjects in the traction group will receive the deneroll extension traction. The subjects will be asked to lie supine on the ground with their legs straight, upper arms by their sides and forearms gently folded across their trunk. The therapist will place the apex of the denneroll either in the mid cervical region or the lower cervical region depending on the apex of cervical curvature deformity of each subject. Initially, participants begin with three minutes of sustained denneroll extension traction and progressed to the goal of 20 min per session with one to two additional minutes per session
  Other Names: Denneroll extension traction

SUMMARY:
Objective: To investigate the immediate and long-term effects of cervical lordosis restoration and anterior head translation (AHT) correction, on pain, disability, autonomic nervous system function and cervical sensorimotor control in Athletes with Chronic nonspecific neck pain.

Methods: 110 (51 female) chronic nonspecific neck patients with a defined hypolordotic cervical spine and AHT posture will be randomly assigned to the control or an experimental group. Both groups will receive a multi-modal program; additionally, the experimental group will receive the denneroll™ cervical traction. Interventions will be applied 3 x per week for 10 weeks. Outcome measures will include absolute rotatory angle (ARA), AHT, neck disability index (NDI), pain intensity, smooth pursuit neck torsion test (SPENT), overall stability index , left and right rotation repositioning accuracy , amplitude and latency of skin sympathetic response . Measures will be assessed at three time intervals: baseline, after 10 weeks of intervention, and at 1-year follow up.

DETAILED DESCRIPTION:
The study is a randomized, single-blind trial. Measurements will be obtained before the randomization, after the intervention period of 10 weeks, and at 12 months. Recruitment will begin following institutional review board approval. The patients will participate in the study after signing an informed consent form prior to data collection. Patients will be included if they were 18 years of age or over; had chronic neck pain (i.e. of more than 3 months duration[19] ; able to attend a full course of 30 treatments, given three times a week. Cervical lordosis measurements (absolute rotation angle ARA C2-C7 using the angle of intersection of two lines drawn along the posterior vertebral body margins of C2 and C7, respectively) were used as a screen for participants' inclusion. [20][21][22] The anterior head translation (AHT) was measured from the posterior superior body of C2 to the vertical line passing through the posterior inferior body of C7. AHT distance had to exceed 25 mm and ARA C2-C7 had to be less than 20° [20] for subjects to be included. Participants were excluded if they presented with any of the following: (i) signs or symptoms of systemic pathology and inflammatory joint disease; (ii) prior history of cervical spine trauma and musculoskeletal system surgery, or disorders related to the spine and extremities. An independent person will assign participants at random to a traditional (control) treatment group (55) or to the intervention group (55). A random number generator was used to select numbers from sealed envelopes. Randomization was conducted through permuted blocks of diverse sizes. These blocks were used to generate a sequence of successively numbered, opaque, sealed envelopes that were kept in a locked drawer. The next envelope in the sequence will be opened by the researcher in the presence of the participant.

Both the intervention group and the traditional treatment group will complete a multimodal program of 10 weeks consisting of myofascial release, thoracic spine mobilization and manipulations, and physical pain relief methods. Additionally, the intervention group will receive the denneroll cervical traction orthotic in an attempt to improve the altered sagittal cervical spine alignment (AHT and ARA C2-C7). The first follow up evaluations will be conducted at the end of the 10-weeks (30 sessions) multimodal program while the second follow up was conducted 1 year after finishing the 10-weeks intervention program.

P All the intervention program will be delivered individually by the same physiotherapist, who has received certified training in these manual techniques in order to minimize inter-therapist variation and enhance fidelity.

ELIGIBILITY:
Inclusion Criteria:

* chronic neck pain (i.e. of more than 3 months duration)
* AHT distance more than 25 mm .
* ARA C2-C7 less than 20°

Exclusion Criteria:

* signs or symptoms of systemic pathology .
* inflammatory joint disease.
* prior history of cervical spine trauma and musculoskeletal system surgery.
* disorders related to the spine and extremities.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-09-05 (Estimated); Study Completion 2021-09-05 (Estimated)

PRIMARY OUTCOMES:
Changes in radiographic measures of cervical alignment | Measures will be assessed at three time intervals: baseline, after 10 weeks of intervention, and at 1-year follow up
  ARA C2-C7 is the angle of intersection of two lines drawn along the posterior vertebral body margins of C2 and C7, respectively) The anterior head translation (AHT) was measured from the posterior superior body of C2 to the vertical line passing through the posterior inferior body of C7.

SECONDARY OUTCOMES:
Changes in Neck disability index | Measures will be assessed at three time intervals: baseline, after 10 weeks of intervention, and at 1-year follow up
  Neck disability index consists of 10 items inquiring about standard daily activities. The responsiveness to change, construct validity, and reliability have been adequately investigated in a variety of patient populations The test can be interpreted as a raw score, with a maximum score of 50.A higher score indicates more patient-rated disability
Changes Numerical pain scale | Measures will be assessed at three time intervals: baseline, after 10 weeks of intervention, and at 1-year follow up
  Neck pain average intensity over the past week was assessed using a number scale from 0-10 with higher scores indicating greater pain intensity.
changes in Cervical joint position sense testing | Measures will be assessed at three time intervals: baseline, after 10 weeks of intervention, and at 1-year follow up
  Assessment of head repositioning accuracy (HRA) with a cervical range of motion (CROM) device will be done according to existing investigations . Participants will be placed in upright neutral seated posture on a stool with no back rest with their feet touching the ground; where their perceived natural head position (NHP) was determined and used as the reference neutral point. The CROM device will be positioned to 0, 0, 0 for x, y, and z rotational displacements. With their eyes closed, participants will be asked to remember their NHP as the starting posture, and then actively rotate their head 30° to the left about the vertical y-axis and then reposition their head back the NHP
Changes in Head and eye motor control | Measures will be assessed at three time intervals: baseline, after 10 weeks of intervention, and at 1-year follow up
  The smooth pursuit neck torsion test (SPNT) will be administered using an Electro-oculography device, to quantify any alteration and improvement in visual motor control

CONTACTS AND LOCATIONS:
Overall Officials: Amina amalmarzouqi, prof, Study Chair — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moustafa I, Youssef ASA, Ahbouch A, Harrison D. Demonstration of Autonomic Nervous Function and Cervical Sensorimotor Control After Cervical Lordosis Rehabilitation: A Randomized Controlled Trial. J Athl Train. 2021 Apr 1;56(4):427-436. doi: 10.4085/1062-6050-0481.19. PMID 33543266